CLINICAL TRIAL: NCT04091295
Title: BLESSED: Expanded Access for DNG64 for Advanced Pancreatic Cancer, Sarcoma and Carcinoma of Breast
Status: Available | Type: Expanded Access
Sponsor: Aveni Foundation (Other)
Responsible Party: Principal Investigator, Erlinda M Gordon, Chief Medical Officer, Aveni Foundation
Other Study IDs: AF19-200
Record Dates: First submitted 2019-08-08; First posted 2019-09-16 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer; Osteosarcoma; MPNST (Malignant Peripheral Nerve Sheath Tumor); Chondrosarcoma; Soft Tissue Sarcoma; Chordoma; Sarcoma; Carcinoma of Breast
Keywords: tumor targeted gene therapy; human cyclin G1 inhibitor; cell cycle control; CCNG1 inhibitor
MeSH Terms: conditions — Pancreatic Neoplasms; Osteosarcoma; Neurofibrosarcoma; Chondrosarcoma; Sarcoma; Chordoma; Breast Neoplasms

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: DNG64 — Intravenous infusions of DNG64 for treatment of advanced pancreatic cancer, sarcoma and carcinoma of breast
  Other Names: DNG64 Chimeric Amphotroopic RNA Vector Encoding a Cyclin G1 Inhibitor

SUMMARY:
Forty patients with pancreatic cancer, sarcoma and carcinoma of breast will receive DNG64 intravenously at a dose of 1-4 x 10e11 colony forming units (cfu) or equivalent 1.0-6.0 x 10e10 RV copies per dose one to three times a week. DNG64 may be given alone or with one or more FDA approved cancer therapies/immunotherapies.

Based on previous Phase 1/2 US based clinical studies, DNG64 does not suppress the bone marrow or cause organ dysfunction, and enhanced immune cell trafficking in tumors may cause the tumors to appear larger or new lesions to appear on CT, PET or MRI. Further, tumor stabilization/regression/remission may occur later during the treatment period. Therefore, DNG64 will be continued regardless of CT, PET or MRI results if the patient has clinical benefit and does not have symptomatic disease progression.

DETAILED DESCRIPTION:
DNG64 is a targeted tumor agnostic gene therapy that displays a Sig-binding peptide for binding to abnormal collagenous Signature (Sig) proteins in the tumor microenvironment and encoding a CCNG1 inhibitor gene for killing cancer cells, its blood supply and stroma producing fibroblasts, thus reducing extracellular matrix production and augmenting drug entry and immune cell trafficking in tumor microenvironment. Enhanced CCNG1 expression has been found in all cancer types tested at the Cancer Center of Southern California as of June 2023. Hence, in July 2023, the USFDA authorized the use of DNG64 as platform therapy upon which one or more FDA approved cancer drugs/ immunotherapies may be added. This would allow a personalized approach in the treatment of all cancer patients.

Forty patients with pancreatic cancer, sarcoma and carcinoma of breast will receive DNG64 intravenously at a dose of 1-4 x 10e11 colony forming units (cfu) or equivalent 1.0-6.0 x 10e10 RV copies per dose one-three times a week. DNG64 may be given alone or with an FDA approved cancer therapy/immunotherapy on physician discretion.

Based on previous Phase 1/2 US based clinical studies, DNG64 does not suppress the bone marrow or cause serious organ dysfunction, and enhanced immune cell trafficking in tumors may cause the tumors to appear larger or new lesions to appear on CT, PET or MRI. Further, tumor stabilization/regression/remission may occur later during the treatment period. Therefore, DNG64 will be continued regardless of CT, PET or MRI results if the patient has clinical benefit and does not have symptomatic disease progression.

If the patient develops a treatment-related >Grade 3 adverse event, the DNG64 infusions will be held and the patient will be monitored until the toxicity has resolved to <Grade 1, and the patient is stable, after which treatment may be resumed. If the adverse event does not resolve to <Grade 1 within 3 weeks, the DNG64 treatment will be held until the data are discussed with the Food and Drug Administration and a decision is made whether to continue or terminate the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥12 years of age, either male or female for patients with sarcoma; >18 years of age, either male or female.with pancreatic cancer or carcinoma of breast.
* Patient has pancreatic cancer or sarcoma or carcinoma of breast confirmed by pathologic examination at diagnosis.
* Patients with advanced metastatic pancreatic cancer who have received systemic therapies such as FOLFIRINOX and gemcitabine + albumin-bound paclitaxel; patients with metastatic sarcoma who have disease progression after two or more lines of systemic treatments and not amenable to surgical resection or radiotherapy; specifically for osteosarcoma: have disease progression after high dose methotrexate, cisplatinum, doxorubicin and ifosfamide; for soft tissue sarcoma: have disease progression after doxorubicin + ifosfamide/mesna, gemcitabine, docetaxel, dacarbazine, trabectedin, pazopanib, eribulin; patients with metastatic carcinoma of breast who have disease progression with standard therapy (ACT), targeted therapies including aromatase inhibitors, trastuzumab, pertuzumab, enhertu, tyrosine kinase inhibitors, immune checkpoint inhibitors; patient who is intolerant to or declines available therapeutic options after documentation that patient has been informed of the available therapeutic options.
* Patient is able to understand or is willing to sign a written informed consent.
* Patient agrees to use barrier contraception during vector infusion period and for 6 weeks after infusion

Exclusion Criteria:

* Patient is unwilling to provide formal informed consent.
* Patient is unwilling to use barrier contraception during vector infusion period and for 6 weeks after infusion

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: ERLINDA M GORDON, MD, Principal Investigator — Sarcoma Oncology Research Center, LLC
Locations (1):
- Sarcoma Oncology Research Center, LLC, Santa Monica, California, United States

REFERENCES:
- [Background] Chawla SP, Chawla NS, Quon D, Chua-Alcala V, Blackwelder WC, Hall FL and Gordon EM: An advanced phase 1/2 study using an XC-targeted gene therapy vector for chemotherapy resistant sarcoma. Sarcoma Res Int 3: 1024, 2016
- [Background] Gordon EM, Hall FL. Rexin-G, a targeted genetic medicine for cancer. Expert Opin Biol Ther. 2010 May;10(5):819-32. doi: 10.1517/14712598.2010.481666. PMID 20384524
- [Background] Chawla SP, Chua VS, Fernandez L, Quon D, Saralou A, Blackwelder WC, Hall FL, Gordon EM. Phase I/II and phase II studies of targeted gene delivery in vivo: intravenous Rexin-G for chemotherapy-resistant sarcoma and osteosarcoma. Mol Ther. 2009 Sep;17(9):1651-7. doi: 10.1038/mt.2009.126. Epub 2009 Jun 16. PMID 19532136
- [Background] Chawla SP, Bruckner H, Morse MA, Assudani N, Hall FL, Gordon EM. A Phase I-II Study Using Rexin-G Tumor-Targeted Retrovector Encoding a Dominant-Negative Cyclin G1 Inhibitor for Advanced Pancreatic Cancer. Mol Ther Oncolytics. 2018 Dec 14;12:56-67. doi: 10.1016/j.omto.2018.12.005. eCollection 2019 Mar 29. PMID 30705966
- [Background] Al-Shihabi A, Chawla SP, Hall FL, Gordon EM. Exploiting Oncogenic Drivers along the CCNG1 Pathway for Cancer Therapy and Gene Therapy. Mol Ther Oncolytics. 2018 Dec 12;11:122-126. doi: 10.1016/j.omto.2018.11.002. eCollection 2018 Dec 21. No abstract available. PMID 30581985
- [Background] Bruckner HW, Chawla SP, Omelchenko N, Brigham DA, Gordon EM. Phase I-II study using DeltaRex-G, a tumor-targeted retrovector encoding a cyclin G1 inhibitor for metastatic carcinoma of breast. Front Mol Med. 2023 May 18;3:1105680. doi: 10.3389/fmmed.2023.1105680. eCollection 2023. PMID 39086675
- [Background] Chawla SP, Olevsky O, Iyengar G, Brigham DA, Omelchenko N, Thomas S, Suryamohan K, Foshag L, Hall FL, Gordon EM. Early-stage CCNG1+ HR+ HER2+ Invasive Breast Carcinoma in Older Women: Current Treatment and Future Perspectives for DeltaRex-G, a CCNG1 Inhibitor. Anticancer Res. 2023 Jun;43(6):2383-2391. doi: 10.21873/anticanres.16406. PMID 37247916
- [Result] Kim S, Federman N, Gordon EM, Hall FL, Chawla SP. Rexin-G(R), a tumor-targeted retrovector for malignant peripheral nerve sheath tumor: A case report. Mol Clin Oncol. 2017 Jun;6(6):861-865. doi: 10.3892/mco.2017.1231. Epub 2017 Apr 28. PMID 28588778